CLINICAL TRIAL: NCT01450059
Title: Maternal-fetal CD4 Microchimerism in HiV Exposed Newborns After Spontaneous Delivery and Cesarean Section
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Horst Buxmann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: 31082011 FRA Mat Fet Chim
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; Microchimerism; Maternal-Fetal Exchange; Gestation; HiV-vertical transmission
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Umbilical Cord blood Blood from peripheral vene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spontaneous delivery: Approximately 15 HiV exposed Newborns with low HiV transmission risk, born via spontaneous delivery.
- Cesarean section: Approximately 15 HiV exposed Newborns with low HiV transmission risk, born via cesarean section.

SUMMARY:
The aim of this single centre study is to measure maternal CD4+ t-cells in HiV exposed Newborns after spontaneous birth in comparison to cesarean section.

This may have an influence on the risk of vertical HiV transmission.

DETAILED DESCRIPTION:
At birth maternal CD4+ t-cells from umbilical cord blood and placenta blood are measured by microchimerism-analysis.

After 6 weeks the maternal CD4+ t-cells are measured in the blood of the babies blood.

Additionally we look for HiV in maternal CD4+ t-cells.

ELIGIBILITY:
Inclusion Criteria:

• HiV exposed Newborns with normal risk of HiV transmission.

Exclusion Criteria:

* HiV exposed Newborns wiht elevated or high risk of HiV transmission.
* HiV exposed Newborns of mothers not full of age.
* missing informed consent of at least the mother
* Outborns
* Asphyxia
* Major congenital defects
* Chromosomal anomalies

Ages: 1 Minute to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 30 HiV exposed newborns born via spontaneuous delivery or cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maternal CD4+ t-cells in HiV exposed Newborns | Six weeks after date of birth
  The maternal CD4+ t-cells are measured by microchimersimanalysis

SECONDARY OUTCOMES:
HiV transmission rate | 6 month after birth
  Measurement of HiV PCR at the age of 6 month after birth
Analysis of HiV in maternal CD4+ t-cells | 2 month after delivery
  HiV-PCR analysis from maternal CD4+ cells
Measurement of maternal CD8+ t-cells in the Newborn | 6 weeks
  Measurement of maternal CD8+ t-cells by microchimerismanalysis

CONTACTS AND LOCATIONS:
Overall Officials: Horst Buxmann, Dr. med., Principal Investigator — Johann Wolfgang Goethe University Hospital Frankfurt/Main, Department of Neonatology
Locations (1):
- Clinic of the Johann Wolfgang-Goethe Univeristy, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] European Collaborative Study; Boer K, England K, Godfried MH, Thorne C. Mode of delivery in HIV-infected pregnant women and prevention of mother-to-child transmission: changing practices in Western Europe. HIV Med. 2010 Jul 1;11(6):368-78. doi: 10.1111/j.1468-1293.2009.00800.x. Epub 2010 Jan 4. PMID 20059573
- [Background] Gemeinsame Erklarung* der Deutschen AIDS-Gesellschaft (DAIG); Osterreichischen AIDS-Gesellschaft (OAG); Kompetenznetzes HIV/AIDS sowie des Robert-Koch-Institutes Berlin (RKI); Deutschen Arbeitsgemeinschaft niederniedergelassener Arzte in der Versorgung von HIV-und AIDS-Patienten (DAGNA); Deutschen Gesellschaft fur Kinderheilkunde und Jugendmedizin (DGKJ); Padiatrischen Arbeitsgemeinschaft AIDS Deutschland (PAAD); Deutschen Gesellschaft fur Gynakologie und Geburtshilfe (DGGG); Nationalen Referenzzentrums fur Retroviren (NRZ) der Deutschen AIDS-Hilfe (DAH). [German-Austrian recommendations for HIV treatment during pregnancy and for newborns exposed to HIV--Update 2008]. Dtsch Med Wochenschr. 2009 Jan;134 Suppl 1:S40-54. doi: 10.1055/s-0028-1123974. Epub 2009 Jan 26. No abstract available. German. PMID 19172555
- [Background] Willasch A, Schneider G, Reincke BS, Shayegi N, Kreyenberg H, Kuci S, Weber G, Van Der Reijden B, Niethammer D, Klingebiel T, Bader P. Sequence polymorphism systems for quantitative real-time polymerase chain reaction to characterize hematopoietic chimerism-high informativity and sensitivity as well as excellent reproducibility and precision of measurement. Lab Hematol. 2007;13(3):73-84. PMID 17984038